CLINICAL TRIAL: NCT04260347
Title: Safe Implementation of Treatments in Stroke (SITS) - Intravenous Thrombolysis in Acute Ischaemic Stroke Patients Over 80 Years, SITS-IVT>80 Years Study
Brief Title: SITS-IVT in Patients >80 Years Study
Acronym: SITS_ELDERLY
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0135-0344
Record Dates: First submitted 2020-01-31; First posted 2020-02-07 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Ischaemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Actilyse® (alteplase) pre-approval
  Interventions: Drug: Alteplase
- Actilyse® (alteplase) post-approval
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Alteplase — Intravenous injection
  Other Names: Actilyse®

SUMMARY:
A non-interventional post-approval study on Safe Implementation of Treatment in Stroke - International Stroke Thrombolysis Register (SITS-ISTR) existing data of intravenous recombinant tissue plasminogen Activator (rt-PA) (0.9 mg/kg) in acute ischaemic stroke patients over 80 years, treated according to the Summary of Product Characteristics (SmPC) in European countries.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 80 years old presenting with acute ischaemic stroke symptoms for which thrombolysis treatment was initiated within 4.5 hours after stroke onset according to SmPC are included.
* Patients over 80 years who received thrombolysis according to SmPC for acute ischaemic stroke (AIS) within 4.5 hours after stroke onset during the period (approximately 3 years) prior to July 2018 are included.

Exclusion Criteria:

* Contraindication(s) to the use of IV thrombolysis per local SmPC.
* Documentation that the patient was enrolled or is planned to be enrolled in an investigational clinical trial at the time of the onset of index event and for the duration of the data collection.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 80 years old presenting with acute ischaemic stroke (AIS) symptoms for which thrombolysis treatment was initiated within 4.5 hours after stroke onset according to the SmPC.
Sampling Method: Probability Sample
Enrollment: 1655 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Observational retrospective study based on existing data collected from the Safe Implementation of Treatment in Stroke-International Stroke Treatment Registry (SITS-ISTR) of ischaemic stroke patients older than 80 years of age treated with Actilyse® (alteplase) according to the Summary of Product Characteristics (SmPC) criteria during post-approval and pre-approval periods.
Pre-assignment Details: The patients were selected based on the sites fulfilling the criteria defined and treated according to the Summary of Product Characteristics (SmPC) of Actilyse® (alteplase) during pre-approval and post-approval period. The data was collected between June 2015 and December 2021. A patient was excluded from the entire cohort when had missing data on one of the selection steps.
Groups:
- Actilyse® (Alteplase) Pre-approval: Patients older than 80 years presenting acute ischaemic stroke symptoms, between June 2015 and July 2018 (or the exact approval date), received once intravenous thrombolysis treatment with off-label Actilyse® (alteplase) within 4.5 hours after stroke onset, according to the Summary of Product Characteristics (SmPC). The recommended total dose was 0.9 milligrams (mg) alteplase per kilogram body weight (maximum of 90 mg) starting with 10% of the total dose as an initial intravenous bolus, immediately followed by the remainder of the total dose infused intravenously over 60 minutes.
- Actilyse® (Alteplase) Post-approval: Patients older than 80 years old presenting acute ischaemic stroke symptoms, between 1st July 2018 (or the first day of the next month after exact approval date) to December 2021, received once intravenous thrombolysis treatment with Actilyse® (alteplase) within 4.5 hours after stroke onset, according to the Summary of Product Characteristics (SmPC). The recommended total dose was 0.9 milligrams (mg) alteplase per kilogram body weight (maximum of 90 mg) starting with 10% of the total dose as an initial intravenous bolus, immediately followed by the remainder of the total dose infused intravenously over 60 minutes.
Period: Overall Study
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Started | 993 | 662
Propensity Score-matched Population | 614 | 614
Completed | 993 | 662
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Propensity score (PS) matched population based on the variables: age, sex, pre-stroke Modified Rankin Scale (mRS) score, baseline National Institute of Health Stroke Scale, systolic blood pressure, glucose level, anti-platelet treatment at stroke onset, hypertension, diabetes, atrial fibrillation, hyperlipidaemia, smoking, previous stroke earlier than 3 months, stroke onset to intravenous thrombolysis treatment start time.
Groups:
- Total: Total of all reporting groups
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval | Total
Number analyzed (Participants) | 614 | 614 | 1228
Age, Continuous [Mean (Standard Deviation); unit: Years] | 86.6 (4.1) | 86.6 (4.3) | 86.6 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 377 | 374 | 751
  Male | 237 | 240 | 477
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic Intracerebral Haemorrhage (SICH) Per Safe Implementation of Thrombolysis - Stroke-Monitoring Study (SITS-MOST) Definition
Description: Defined as the number of participants presenting intracerebral haemorrhage (parenchymatous haemorrhage type 2, PH2), at the 22-36 hours post-treatment scan or earlier, if clinically indicated, combined with neurological deterioration leading to an increase of 4 points on the National Institutes of Health Stroke Scale (NIHSS) from baseline to 24h or death within 24 hours (SITS-MOST definition). The NIHSS is a neurological examination tool used to objectively quantify stroke severity. It is composed by 11 items, 3 of which with more than one component, scoring between 0 (normal function) and 2, 3, 7 or 8 (highest degree of impairment) for a specific ability (item). The sum of the individual scores from each item originate the total NIHSS score, where: 0 = no stroke symptoms; 1-4 = minor stroke; 5-15 = moderate stroke; 16-20 = moderate to severe stroke; and 21-42 = severe stroke.
Time Frame: Up to 36 hours after stroke onset, between June 2015 and December 2021
Population: Propensity score matched population based on the variables: age, sex, pre-stroke Modified Rankin Scale score, baseline National Institute of Health Stroke Scale, systolic blood pressure, glucose level, anti-platelet treatment at stroke onset, hypertension, diabetes, atrial fibrillation, hyperlipidaemia, smoking, previous stroke earlier than 3 months, stroke onset to intravenous thrombolysis treatment start time. Participants with missing values were excluded from the analysis of this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Number analyzed (Participants) | 599 | 603
Participants | 14 | 15
Statistical Analysis 1: Comparison: Actilyse® (Alteplase) Pre-approval vs Actilyse® (Alteplase) Post-approval; Test type: Other; p = 1.000, Chi-squared; Risk Ratio (RR) = 1.064, 95% CI 2-sided [0.345 to 1.784] — Actilyse® (alteplase) pre-approval participants were used as reference group

2. Primary Outcome: Mortality Within 90 Days, Defined as the Number of Participants With a Death Event
Description: Number of participants who died within 90 days as classified by the investigator according to cause: cerebral infarct, cerebral haemorrhage, cerebral infarct and haemorrhage unspecified, myocardial infarct, pulmonary embolism, pneumonia, other vascular cause, unknown and other cause of death. The International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) was used.
Time Frame: Up to 90 days after stroke onset, between June 2015 and December 2021
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Number analyzed (Participants) | 566 | 589
Participants | 161 | 149
Statistical Analysis 1: Comparison: Actilyse® (Alteplase) Pre-approval vs Actilyse® (Alteplase) Post-approval; Test type: Other; p = 0.254, Chi-squared; Risk Ratio (RR) = 0.889, 95% CI 2-sided [0.699 to 1.08] — Actilyse® (alteplase) pre-approval participants were used as reference group

3. Primary Outcome: Functional Independency, as Defined by a mRS (Modified Rankin Score) 0-2 Within 90 Days
Description: Defined as the number of participants classified with a modified Rankin score (mRS) of 0, 1 or 2 within 90 days. The mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke. The score has a scale from 0 to 6, where: 0 = no symptoms at all; 1 = no significant disability despite symptoms, able to carry out all usual duties and activities; 2 = slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance; 3 = moderate disability, requiring some help but able to walk without assistance; 4 = moderately severe disability, unable to walk without assistance and unable to attend own bodily needs without assistance; 5 = severe disability, bedridden, incontinent and requiring constant nursing care and attention; and 6 = dead.
Time Frame: Up to 90 days after stroke onset, between June 2015 and December 2021
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Number analyzed (Participants) | 554 | 578
Participants | 205 | 233
Statistical Analysis 1: Comparison: Actilyse® (Alteplase) Pre-approval vs Actilyse® (Alteplase) Post-approval; Test type: Other; p = 0.280, Chi-squared; Risk Ratio (RR) = 1.089, 95% CI 2-sided [0.942 to 1.237] — Actilyse® (alteplase) pre-approval participants were used as reference group

4. Secondary Outcome: Stroke Severity, Defined by the National Institute of Health's Stroke Scale (NIHSS)
Description: Defined by the total National Institutes of Health Stroke Scale (NIHSS) score presented by the participants of each group at baseline. The NIHSS is a neurological examination tool used to objectively quantify stroke severity. It is composed by 11 items, 3 of which with more than one component, scoring between 0 (normal function) and 2, 3, 7 or 8 (highest degree of impairment) for a specific ability (item). The sum of the individual scores from each item originate the total NIHSS score, where: 0 = no stroke symptoms; 1-4 = minor stroke; 5-15 = moderate stroke; 16-20 = moderate to severe stroke; and 21-42 = severe stroke.
Time Frame: At baseline, defined as the ischaemic stroke hospital admission date, between June 2015 and December 2021
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Number analyzed (Participants) | 614 | 614
Units on a scale | 10.5 [7 to 16] | 11 [6 to 17]
Statistical Analysis 1: Comparison: Actilyse® (Alteplase) Pre-approval vs Actilyse® (Alteplase) Post-approval; Test type: Other; p = 0.916, Wilcoxon (Mann-Whitney); Standardized Mean Difference (SMD) = 0.016, 95% CI 2-sided [-0.096 to 0.128] — SMD = Difference in the mean between groups / Standard deviation Actilyse® (alteplase) pre-approval participants were used as reference group

5. Secondary Outcome: Number of Participants With a Modified Rankin Score (mRS) of 0-1 Within 90 Days
Description: Defined as the number of participants achieving of a modified Rankin score (mRS) of 0 or 1 within 90 days. The mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke. The score has a scale from 0 to 6, where: 0 = no symptoms at all; 1 = no significant disability despite symptoms, able to carry out all usual duties and activities; 2 = slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance; 3 = moderate disability, requiring some help but able to walk without assistance; 4 = moderately severe disability, unable to walk without assistance and unable to attend own bodily needs without assistance; 5 = severe disability, bedridden, incontinent and requiring constant nursing care and attention; and 6 = dead.
Time Frame: Up to 90 days after stroke onset, between June 2015 and December 2021
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Number analyzed (Participants) | 554 | 578
Participants | 142 | 158
Statistical Analysis 1: Comparison: Actilyse® (Alteplase) Pre-approval vs Actilyse® (Alteplase) Post-approval; Test type: Other; p = 0.561, Chi-squared; Risk Ratio (RR) = 1.066, 95% CI 2-sided [0.872 to 1.261] — Actilyse® (alteplase) pre-approval participants were used as reference group

6. Secondary Outcome: Number of Participants With Symptomatic Intracerebral Haemorrhage (SICH) Per European Cooperative Acute Stroke Study 2 (ECASS 2) Definition
Description: Defined as the number of participants with any intracerebral haemorrhage including haemorrhagic infarctions at the 22-36 hours post-treatment scan combined with neurological deterioration leading to an increase of 4 points on the National Institutes of Health Stroke Scale (NIHSS) or death within 7 days. The NIHSS is a neurological examination tool used to objectively quantify stroke severity.It is composed by 11 items, 3 of which with more than one component, scoring between 0 (normal function) and 2, 3, 7 or 8 (highest degree of impairment) for a specific ability (item). The sum of the individual scores from each item originate the total NIHSS score, where: 0 = no stroke symptoms; 1-4 = minor stroke; 5-15 = moderate stroke; 16-20 = moderate to severe stroke; and 21-42 = severe stroke.
Time Frame: Up to 7 days after stroke onset, between June 2015 and December 2021
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Number analyzed (Participants) | 594 | 603
Participants | 24 | 30
Statistical Analysis 1: Comparison: Actilyse® (Alteplase) Pre-approval vs Actilyse® (Alteplase) Post-approval; Test type: Other; p = 0.522, Chi-squared; Risk Ratio (RR) = 1.231, 95% CI 2-sided [0.707 to 1.756] — Actilyse® (alteplase) pre-approval participants were used as reference group

7. Secondary Outcome: Time From Onset of Symptoms to Start of Intravenous Thrombolysis (IVT) Treatment
Description: Time in minutes from the onset of ischaemic stroke symptoms to start of treatment with intravenous thrombolysis with Actilyse® (alteplase).
Time Frame: Up to 4.5 hours after stroke onset, between June 2015 and December 2021
Population: Propensity score matched population based on the variables: age, sex, pre-stroke Modified Rankin Scale score, baseline National Institute of Health Stroke Scale, systolic blood pressure, glucose level, anti-platelet treatment at stroke onset, hypertension, diabetes, atrial fibrillation, hyperlipidaemia, smoking, previous stroke earlier than 3 months, stroke onset to intravenous thrombolysis treatment start time.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Number analyzed (Participants) | 614 | 614
Minutes | 153 [111.25 to 195] | 151 [114.25 to 195]
Statistical Analysis 1: Comparison: Actilyse® (Alteplase) Pre-approval vs Actilyse® (Alteplase) Post-approval; Test type: Other; p = 0.810, Wilcoxon (Mann-Whitney); Standardized Mean Difference (SMD) = -0.021, 95% CI 2-sided [-0.133 to 0.091] — SMD = Difference in mean between groups / Standard deviation Actilyse® (alteplase) pre-approval participants were used as reference group

8. Secondary Outcome: Time From Onset of Symptoms to Door (or Captured in the Registry Arrival at the Hospital)
Description: Time in minutes from the onset of ischaemic stroke symptoms to hospital door or the registry arrival at the hospital.
Time Frame: Up to 4.5 hours after stroke onset, between June 2015 and December 2021
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Number analyzed (Participants) | 614 | 614
Minutes | 93 [65 to 135] | 88 [62 to 128]
Statistical Analysis 1: Comparison: Actilyse® (Alteplase) Pre-approval vs Actilyse® (Alteplase) Post-approval; Test type: Other; p = 0.179, Wilcoxon (Mann-Whitney); Standardized Mean Difference (SMD) = -0.085, 95% CI 2-sided [-0.199 to 0.03] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Door to Needle Time
Description: Time in minutes from hospital door or registry arrival at the hospital to start of treatment with intravenous thrombolysis (IVT) with Actilyse® (alteplase)
Time Frame: Up to 4.5 hours after stroke onset, between June 2015 and December 2021
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
Number analyzed (Participants) | 614 | 614
Minutes | 46 [27 to 75] | 48 [30 to 79]
Statistical Analysis 1: Comparison: Actilyse® (Alteplase) Pre-approval vs Actilyse® (Alteplase) Post-approval; Test type: Other; p = 0.275, Wilcoxon (Mann-Whitney); Standardized Mean Difference (SMD) = 0.042, 95% CI 2-sided [-0.072 to 0.156] — [estimate comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: As this is a study with secondary use of data retrieved from Safe Implementation of Treatment in Stroke-International Stroke Treatment Registry (SITS-ISTR), safety monitoring/reporting on an individual case level is not applicable. All-Cause Mortality, Serious Adverse Events and Other Adverse Events are not collected in the database. "0" total Number of Participants at Risk means "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Actilyse® (Alteplase) Pre-approval | Actilyse® (Alteplase) Post-approval
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04260347/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04260347/SAP_001.pdf